CLINICAL TRIAL: NCT03243799
Title: Effectiveness of a Psychoeducational Group Intervention Conducted by Primary Health Care Nurses in Patients With Depression and Physical Comorbidity
Brief Title: Effectiveness of a Psychoeducational Group Intervention in Patients With Depression and Physical Comorbidity
Acronym: PsiCoDep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI16/01272
Record Dates: First submitted 2017-07-25; First posted 2017-08-09 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will participate in psychoeducational groups: 12 weekly 90-minute sessions led by two nurses from Primary Care, consisting of health education on chronic physical illness and depressive symptoms.
  Group psychoeducation.
  Interventions: Behavioral: Group psychoeducation
- Control Group (No Intervention): Usual clinical care

INTERVENTIONS:
Behavioral: Group psychoeducation — Educational group sessions for patients with depression and physical comorbidities in order to improve the degree of control of their illnesses
  Arms: Intervention Group

SUMMARY:
The primary aim is to evaluate the effectiveness of an intervention based on a psychoeducational program carried out by primary care nurses, to improve the rate of remission and response of depression in patients with physical chronic illness (diabetes, COPD, asthma and / or ischemic heart disease). Secondarily, to assess the cost-effectiveness of the intervention, the effectiveness to improve the control of physical pathology, the impact on quality of life and the feasibility of the intervention.

Methods: a multicentre, randomized clinical trial, with two groups and 1 year follow-up evaluation. Economic evaluation study. We will study 504 patients (252 in each group), over 50 years assigned to 25 primary care teams (PC) from Catalonia (urban, semi-urban and rural) with major depression and with at least one of the diseases: diabetes mellitus type 2, chronic obstructive pulmonary disease, asthma, and / or ischemic heart disease. They will be distributed randomly into two groups. The intervention group will participate in psychoeducational groups: 12 weekly 90-minute sessions led by two nurses from PC, consisting of health education on chronic physical illness and depressive symptoms.

Main measurements: clinical remission of depression and / or response to intervention (Beck depression inventory: BDI-II). Secondary measures: improvement in control of chronic disease (blood test and physical parameters), drug compliance (test Morinsky-Green and number of packaging), quality of life (EQ-5D), medical service utilization (appointments and hospital admissions due to complications) and feasibility of the intervention (satisfaction and compliance). Evaluations will be masked and conducted at 0, 3 and 12 months. At 6 months, patients will receive a call from nurses.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one of the following diseases: type 2 diabetes mellitus, chronic obstructive pulmonary disease, asthma, and / or ischemic heart disease.
* Meet major depression criteria at the time of the study: Score above 13 on the BDI-II scale.
* Possibility of follow-up of one year by the same primary care team.
* At least read and write Spanish or Catalan.

Exclusion Criteria:

* Diagnosis of dementia or moderate or high cognitive impairment (5 or more errors according to the pfeiffer scale).
* Major depression with psychotic symptoms or with other serious psychiatric comorbidities.
* Moderate or high risk of suicide (6 or more points on the MINI suicide scale).
* Dependency disorders due to alcohol or other drug abuse.
* Advanced stage physical disease.
* Inability to travel to the center.
* Be receiving some psychological therapy by the Center of mental health (CSM) of reference

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in rate of remission of depression | At 12 months of follow-up
  Changes in the score of the BDI-II scale

SECONDARY OUTCOMES:
Changes in rate of remission of depression | At 3 months of follow-up
  Changes in the score of the BDI-II scale
Changes in the control of DM2 | At 12 months of follow-up
  Changes in HbA1c
Changes in the control of COPD | At 12 months of follow-up
  Changes in FEV1
Changes in the control of asthma | At 12 months of follow-up
  Changes in FEV1
Changes in the control of Ischemic heart disease | At 12 months of follow-up
  Changes in LDL cholesterol
Referrals to mental health | At 12 months of follow-up
  Number of visits to mental health centers
Record of therapeutic compliance | At 12 months of follow-up
  Morisky-Green test
Changes in the quality of life | At 12 months of follow-up
  Measured by the EuroQol scale (EQ-5D)
Quantification of the use of services | At 12 months of follow-up
  Number of hospital admissions
Satisfaction with the intervention | At 3 months of follow-up
  Survey at the end of the intervention
Adherence to the intervention | At 3 months of follow-up
  Number of assisted sessions
Qualitative changes of the state of mind at the end of the intervention | At 3 and 12 months of follow-up
  better, equal or worse
Qualitative changes of the state of health at the end of the intervention | At 3 and 12 months of follow-up
  better, equal or worse

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Atenció Primària (CAP) Santa Margarida de Montbui, Santa Margarida de Montbui, Barcelona, Spain

REFERENCES:
- [Derived] Casanas R, Martin Royo J, Fernandez-San-Martin MI, Raya Tena A, Mendioroz J, Sauch Valmana G, Masa-Font R, Casajuana-Closas M, Fernandez Linares EM, Cols-Sagarra C, Gonzalez Tejon S, Foguet-Boreu Q, Martin Lopez LM. Effectiveness of a psychoeducation group intervention conducted by primary healthcare nurses in patients with depression and physical comorbidity: study protocol for a randomized, controlled trial. BMC Health Serv Res. 2019 Jun 26;19(1):427. doi: 10.1186/s12913-019-4198-7. PMID 31242892